CLINICAL TRIAL: NCT03292120
Title: Venous to Arterial Carbon Dioxide Difference (P₍ᵥ-ₐ₎CO₂): Predictor of Septic Patient Prognosis Depending on the ScvO₂
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2016-07; 2016-A00586-45 (Other: n°IDRCB)
Record Dates: First submitted 2017-09-20; First posted 2017-09-25 (Actual); Last update posted 2019-05-08 (Actual); Status verified 2019-05

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with septic shock (Experimental)
  Interventions: Other: measure of the SOFA score

INTERVENTIONS:
Other: measure of the SOFA score — The Sequential Organ Failure Assessment (SOFA) Score predicts ICU mortality based on lab results and clinical data.

SUMMARY:
the investigators will include 120 patients with a diagnosis of septic shock in accordance with the definition given by the 2001 expert consensus. Two groups of patients are likely to participate in this study: Patient hospitalized in intensive care for a septic shock = Primary patient + patient who develops, the waning of his hospitalization in intensive care for another reason, a septic shock = Secondary patient. Haemodynamic monitoring by transpulmonary thermodilution allow a patient's close monitoring during the initial phase supported. The clinical and biological data, demographic and the severity scores are collected for each patient during the first three days of stay. To predict the unfavorable evolution of the patients, a measure of the SOFA score at the input (J0) and third day (J2) is performed. the investigators analyzed mortality at day 28 in patients with increased P₍ᵥ-ₐ₎CO₂ and those with increasing of organ failure. This research will be conducted according to good clinical practice. An information will be distributed to patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a diagnosis of septic shock
* Initial lactate in patients should be≥ 2 mmol / L.
* The presence of circulatory insufficiency defined by a systolic blood pressure ≤ 90 mmHg (or a drop in blood pressure≥ 50 mmHg in hypertensive patients)
* One or more of the following: oliguria defined as diuresis≤ 0,5 mL/ kg / h for at least two hours; the presence of signs of cerebral hypoperfusion; the highlighting of mottling
* The presence of a femoral arterial catheter and a central venous line in the superior vena cava position
* Hemodynamic monitoring with semi-invasive monitoring of cardiac output with thermodilution

Exclusion Criteria:

* Patient no longer in the initial phase of septic shock
* Absence of semi-invasive cardiac monitoring with thermodilution
* Vulnerable people
* Absence of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
measure of the SOFA score | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: jean olivier ARNAUD, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assisitance Publique Hopitaux de Marseille, Marseille, France